CLINICAL TRIAL: NCT01785706
Title: COPD Research Registry
Status: Completed | Type: Observational
Sponsor: COPD Foundation (Other)
Collaborators: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2357
Record Dates: First submitted 2013-01-11; First posted 2013-02-07 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years

SUMMARY:
The COPD Research Registry is a confidential database of individuals diagnosed with COPD or at risk of developing COPD. The Registry was established in 2007 by the COPD Foundation with the purpose of providing a mechanism for researchers to boost enrollment in clinical trials and other research studies. The COPD Foundation is working with National Jewish Health in Denver, Colorado to serve as the Registry's Data Coordinating Center and to ensure strictest confidentiality of participant information.

ELIGIBILITY:
Inclusion Criteria:

-Individuals over the age of 18 who have COPD or may be considered to be at increased risk for development of COPD.

Exclusion Criteria:

-Individuals under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with COPD or at-risk of developing COPD.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2007-03; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The COPD Foundation expects to assist at least 8 researchers (with patient recruitment) annually. | Up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: James Crapo, M.D., Principal Investigator — National Jewish Health
Locations (1):
- COPD Foundation, Miami, Florida, United States